CLINICAL TRIAL: NCT00680394
Title: Comparing Two Regimens for Medical Abortion: Mifepristone+Misoprostol Versus Misoprostol Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol 1.2.1
Record Dates: First submitted 2008-03-03; First posted 2008-05-20 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Pregnancy Termination
Keywords: abortion; medical abortion; mifepristone; misoprostol
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mifepristone+misoprostol (Experimental): 200 mg mifepristone+ 800 mcg buccal misoprostol
  Interventions: Drug: mifepristone; Drug: misoprostol
- misoprostol (Experimental): 800 mcg buccal misoprostol+placebo
  Interventions: Drug: misoprostol; Drug: placebo

INTERVENTIONS:
Drug: mifepristone — 200 mg mifepristone
  Arms: mifepristone+misoprostol
Drug: misoprostol — 800 buccal misoprostol + matching placebo or 1600 buccal misoprostol
Drug: placebo — 800 buccal misoprostol + matching placebo or 1600 buccal misoprostol
  Arms: misoprostol

SUMMARY:
A double blinded, placebo-controlled randomized trial to compare the safety, efficacy and acceptability of two medical abortion regimens up to 63 days' LMP. The first regimen will include a 200 mg oral dose of mifepristone followed by 800 mcg buccal misoprostol. The second regimen will include two 800 mcg doses of buccal misoprostol. We hypthesize that both methods work well, but that the mifepristone regimen will have an efficacy rate of approximately 95%, and misoprostol alone will be closer to 90%. We will consider a greater than 5% difference to be clinically meaningful.

DETAILED DESCRIPTION:
Non-surgical abortion methods have the potential to improve the quality and safety of women's reproductive health in the developing world. However, until recently, widespread availability and utilization of medical abortion with mifepristone in low resource countries has been restricted by the limited availability of mifepristone and perceived high cost of the drug, while the low and varied rates of efficacy of the misoprostol alone regimens have hindered its widespread adoption. In recent years, a handful of new mifepristone and misoprostol products have come to the market, easing the availability and reducing the cost of both drugs, and therefore making their introduction in new settings more feasible. Nonetheless, mifepristone is much more expensive than misoprostol (approximately $4 - 6 a tablet versus $0.35 a tablet) and often a large part of the cost of the medical abortion cost. In this respect, this study provides an important opportunity to better understand the real difference in efficacy of the two regimens in addition to the costs and benefits of these two non-surgical abortion regimens.

The study will contribute greatly to the literature on medical abortion. First, it will be the first randomized trial to compare two buccal regimens (and the second ever to compare mifepristone+misoprostol with misoprostol alone. Second, if proven efficacious, it promises to offer alternative regimens for use in women with gestations up to 63 days' LMP. Third, it may create evidence in support of shortening the time to abortion completion, by offering all women in the mifepristone arm the chance to complete their abortions 24 hours after mifepristone, instead of the standard 48 hours later. Lastly, it provides a unique opportunity to systematically and in a non-biased manner, compare the side effects and acceptability of these two regimens, thereby creating more information to help providers and policy makers debate the relative costs and benefits of these two medical abortion regimens.

A total of 700 women will be recruited. We assume that the efficacy of mifepristone plus buccal misoprostol is approximately 95%. The efficacy of misoprostol alone for medical abortion, via the vaginal route, is 88%. The efficacy of misoprostol alone via the buccal route is not known, nor is the efficacy via the buccal route with repeat dosing after a 24 hour interval. We expect that the efficacy with buccal misoprostol should be similar to that with vaginal misoprostol based on both pharmokinetic and clinical data.

We assume that the efficacy of mifepristone plus buccal misoprostol in our research settings will be 95%. A difference in efficacy of buccal misoprostol alone of at least 5% (90%) is clinically meaningful to providers and women.

Using alpha = 0.05 with a one-sided test and power = 0.80, the number needed to demonstrate this difference is 664 (334 in each arm). Assuming 5% will drop out or not complete the protocol, we plan to enroll a total of 700 women.

The primary endpoint is efficacy; safety, acceptability and side effects will be assessed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 63 days by LMP, ultrasound or clinical assessment.
* General good health including absence of conditions which contraindicate the use of mifepristone and misoprostol for pregnancy termination.
* Agrees to return for follow-up visit and willing to provide an address and/or telephone number for purposes of follow-up.
* Able to consent to study participation.

Exclusion Criteria:

* Gestational age > 63 days
* Confirmed or suspected ectopic or molar pregnancy
* Contraindications to medical abortion including IUD in place (must be removed before procedure), chronic adrenal failure, concurrent long-term corticosteroid therapy, history of allergy to mifepristone, misoprostol or prostaglandin, hemorrhagic disorders or concurrent anticoagulant therapy, inherited porphyries.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Efficacy defined as complete abortion without recourse to surgical abortion. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- La Rabta Hospital, Tunis, Tunisia
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Blum J, Raghavan S, Dabash R, Ngoc Nt, Chelli H, Hajri S, Conkling K, Winikoff B. Comparison of misoprostol-only and combined mifepristone-misoprostol regimens for home-based early medical abortion in Tunisia and Vietnam. Int J Gynaecol Obstet. 2012 Aug;118(2):166-71. doi: 10.1016/j.ijgo.2012.03.039. Epub 2012 Jun 8. PMID 22682768
- [Derived] Ngoc NT, Blum J, Raghavan S, Nga NT, Dabash R, Diop A, Winikoff B. Comparing two early medical abortion regimens: mifepristone+misoprostol vs. misoprostol alone. Contraception. 2011 May;83(5):410-7. doi: 10.1016/j.contraception.2010.09.002. Epub 2010 Oct 18. PMID 21477682